CLINICAL TRIAL: NCT06050811
Title: A Randomised, Placebo-controlled, Double-blinded Crossover Trial Investigating the Effect of a Dietary Prebiotic on Clinical, Metabonomic, Microbiological, and Immunological Outcomes in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: Prebiotics in Reducing Inflammation and Clinical Endpoints in Ulcerative Colitis (PRInCE-UC)
Acronym: PRInCE-UC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Berkshire NHS Foundation Trust (Other Government)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PRInCE-UC
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
Keywords: Gut microbiota; Prebiotic; Human milk oligosaccharide
MeSH Terms: conditions — Colitis, Ulcerative | interventions — 2'-fucosyllactose

STUDY DESIGN:
Intervention Model Description: Volunteers will be assigned randomly to take either prebiotic or placebo during an initial 28 day period. A 21 day wash-out period, during which no prebiotic or placebo will be consumed, will separate the 28 day treatment periods and there will be a further washout at the end (to ascertain the duration of prebiotic effect). There will therefore be four test periods randomly assigned (prebiotic; washout; placebo; washout; OR placebo; washout; prebiotic; washout).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The candidate prebiotic and placebo will be pre-packaged randomly off-site, and the investigator and patient will not know whether the prebiotic or the placebo is being administered. This will be unmasked for the data analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic supplement (Experimental): 5 g 2'-Fucosyllactose per day
  Interventions: Dietary Supplement: 2'-Fucosyllactose
- Placebo (Placebo Comparator): 5 g maltodextrin per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 2'-Fucosyllactose — 2'-Fucosyllactose given orally with water or food for four weeks, followed by a three week washout period.
  Arms: Prebiotic supplement
Dietary Supplement: Placebo — Maltodextrin given orally with water or food for four weeks, followed by a three week washout period.
  Arms: Placebo

SUMMARY:
The community of microbes living in the gut is called the 'gut microbiome'. Changing this could be an exciting new way of treating people living with ulcerative colitis (UC).

UC is a type of inflammatory bowel disease. It affects 4 in every 1000 people in the UK. UC causes severe episodes of inflammation leading to bloody diarrhoea. The gut microbes of people living with UC are different to those in healthy people. This may be part of the reason people with UC have a more inflamed gut.

Prebiotics are types of fibre in the diet which help feed the positive microbes in the colon. Eating them can change the make-up and activity of the bugs which live in our gut in a good way.

The goal of this clinical trial is to test the effect of a type of prebiotic called a human milk oligosaccharide (HMO) on the symptoms of patients with UC. The main questions it aims to answer are:

* Can a prebiotic improve symptoms for patients living with UC?
* Can a prebiotic improve the gut microbiota of people living with UC, and improve markers of inflammation, metabolism and immune function?

Patients will take a sachet containing either the prebiotic or a placebo for four weeks, then swap to the other sachet. The trial will be double-blind and randomised. This 'crossover' design means patients act as their own control, which is important in gut microbiology studies. The prebiotic's effect on patient symptoms, metabolism and immune system will be measured. The investigators plan to recruit 44 participants over 18 months. Their urine, blood and stool will be tested.

This project will be the first 'bench to bedside' study into the use of prebiotics in IBD. The treatment in this project is rooted in gut model studies. Different prebiotics were tested in the lab to determine which was the best to use for the trial. This 'lab first' approach is a first of its kind.

DETAILED DESCRIPTION:
This dietary intervention study will be carried out in a double-blind, cross-over manner, whereby 44 participants with mild to moderately active UC will be asked to consume an appropriate dose of the candidate prebiotic (2'-Fucosyllactose, a human milk oligosaccharide) for 28 days followed by a 28 day feeding period with an equivalent placebo (maltodextrin), or vice versa. Prebiotics are generally available in sachet form and participants will be instructed on how to take them each day.

Volunteer bowel habit, symptom scoring and quality of life: During supplementation and washout periods, the volunteers will be sent questionnaires to record their bowel habit, use of medication and adverse events. Volunteers will record the number of bowel movements per day, Bristol stool scale scores and any symptoms of bloating or abdominal discomfort (rated as none, mild, moderate or severe). Validated scoring systems will be used, namely the Simple Clinical Colitis Activity Index (SCCAI), a marker of clinical activity, and the IBD-Control questionnaire which is the International Consortium for Health Outcomes Measurement measure of choice for assessing disease-specific quality of life in IBD.

Selectivity index: The impact of prebiotic feeding upon relative numbers of potentially health promoting Bifidobacterium, Roseburia, Faecalibacteria and Lactobacilli (beneficial), upon numbers of commensal Eubacterium spp., Atopobium spp. and upon numbers of potentially detrimental members of the gut microflora namely Escherichia coli, proteolytic Bacteroides spp. and the Clostridium perfringens/histolyticum group will be determined within the faecal microflora. Moreover, functional capacity of the microbiome and the impact on the host metabolic phenotype will be determined by 1H-Nuclear Magnetic Resonance (NMR) spectroscopy-based metabonomics. These global profiles contain information relating directly to microbial metabolic processes, trans- genomic interactions as well as host endogenous metabolism. Through application of this top-down systems biology approach, biochemical responses of the host and microbiota to prebiotic exposure can be characterised.

Gut microbiota composition studies: Fluorescent in situ hybridisation (FISH) will be used to identify and enumerate principal anaerobic bacteria in the human studies, and flow cytometry will enable high throughput and sensitivity. In addition, a full qualitative assessment of community structure through a metagenomic approach using high capacity sequencing (454 pyrosequencing or similar) will be applied.

1H-NMR spectroscopy-based metabolic profiling studies: In this proposal, 1H-NMR spectroscopy will be applied to characterise global metabolic signatures from biological samples collected throughout the human trials, using standard one-dimensional NMR experiments. Gut microbiology and metabonomic data will be integrated using data fusion techniques (for example, bidirectional partial least squares multi-block data analysis) to generate mechanistic understanding of system-level changes and optimise extraction of clinically relevant molecular information. It is anticipated that this analysis will provide a measure of how prebiotic based intervention during the clinical trial has affected the human metabonome in a manner closer to 'health.'

Immunological assessments: Blood and faecal specimens will be used to determine immune cell counts and phenotypes. These data will show immunological status of the patients at any particular time of the trial - including inflammatory issues.

Immune cell subsets interacting with antigen presentation cell populations: The investigators will compare antigen-presentation by differentiated cell types (professional and stromal) and the extent to which they interact with effector T-cell subsets. It is likely that initial presentation of antigen to the immune system will differ between these groups and quantifying these interactions using 4-colour fluorescence immunohistology will provide mechanistic information of these processes and the progression of the UC disease state.

Data collected will be bacterial community profiles, immunological markers, blood/serum measurements, volunteer questionnaires, NMR-based metabonomic data, microbial end products and patient symptoms. These data will mostly be numerical and in the form of Excel spreadsheets, but will also include spectra data files, raw sequence files and food diary records (MS word/REDCap). Software for data analysis will be SAS (Statistical Analysis Software). Only the metabonomic NMR spectroscopy and microbial sequencing data files will generate moderately large data volumes. The investigators will identify community standards for data formatting for eventual deposit in data repositories.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Adults (aged from 18 to 64)
* Diagnosis of ulcerative colitis by endoscopy and histology
* Mildly or moderately active UC (based on symptom score and gastroenterologist opinion, with elevated serum C-reactive protein above reference range for local laboratory and/or faecal calprotectin of 150 μg/g or greater and/or endoscopic disease activity, the latter three criteria having been within the past 2 months.)

Exclusion Criteria:

* Patients with acute severe colitis, as defined by the Truelove and Witts criteria
* Intake of an experimental drug within four weeks prior to study
* Former participation in prebiotic or laxative trials within the previous three months
* Use of antibiotics within the previous four weeks
* Introduction of an immunomodulator or advanced therapy (e.g. biologic) within 12 weeks or dose change of an immunomodulator or advanced therapy within 6 weeks
* Introduction of oral 5-ASA within 8 weeks, or dose change of an oral 5-ASA agent within 2 weeks
* Use of corticosteroids within preceding 6 weeks or during trial period
* Intake of other specific prebiotics (such as oligosaccharides e.g. inulin), or probiotics (e.g. live yoghurts, other fermented products), drugs active on gastrointestinal motility, or a laxative of any class, for four weeks prior to study.
* Women who are lactating, pregnant or planning pregnancy during the study period.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Clinical response measured using Simple Clinical Colitis Activity Index | Four weeks
  Clinically significant improvement in patient symptoms as defined by a decrease in Simple Clinical Colitis Activity Index Score of greater than or equal to 2 points from baseline.

SECONDARY OUTCOMES:
Clinical remission measured using Simple Clinical Colitis Activity Index | Four weeks
  Clinical remission as defined by a Simple Clinical Colitis Activity Index Score of less than or equal to 2 points.
Colonic inflammation | Four weeks
  Changes in markers of colonic inflammation such as faecal calprotectin
Changes in faecal microbiota composition | Four weeks
  Faecal microbiota composition before and after intervention or placebo will be assessed quantitatively by a combination of fluorescent in situ hybridisation flow cytometry and 16S rRNA gene sequencing
Faecal bacterial metabolites | Four weeks
  Changes in metabolites such as short chain fatty acids measured using targeted and non-targeted metabolomic techniques
Changes in urinary metabolites | Four weeks
  Changes in concentration of metabolites measured in urine using targeted and non-targeted metabolomic techniques
Changes in serum metabolites | Four weeks
  Changes in concentration of metabolites measured in serum using targeted and non-targeted metabolomic techniques
Stool consistency | Four weeks
  Stool consistency as measured by the Bristol Stool Chart
IBD-related quality of life assessed by IBD Control score | Four weeks
  IBD-related quality of life as measured by change in Inflammatory Bowel Disease Control score, measured on a scale of 0 to 16, with 16 being the maximum score representing the best quality of life, and 0 being the minimum score.
Host immune system changes | Four weeks
  Immune cell counts using fluorescence immunohistology

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Gibson, PhD, Study Director — University of Reading
Locations (1):
- Royal Berkshire NHS Foundation Trust, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
On completion of the project anonymised experimental data and relevant metadata will be deposited in the University of Reading Research Data Archive for long-term preservation and made available under open licence for re-use by the scientific community. It is envisaged that relevant data will be available 6 months following the end of the project and no later than publication of related findings.